CLINICAL TRIAL: NCT07160335
Title: A Multicenter, Randomized, Double-Blind, Parallel-Controlled Phase I Clinical Study to Evaluate the Pharmacokinetic Profile, Efficacy, Safety and Immunogenicity of HLX17 vs. Keytruda® (US-sourced Keytruda®) in Multiple Resected Solid Tumors
Brief Title: A Phase I Clinical Study to Evaluate the PK Profile, Efficacy, Safety and Immunogenicity of HLX17 vs. Keytruda® in Multiple Resected Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX17-MRST001
Record Dates: First submitted 2025-08-22; First posted 2025-09-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer; Melanoma; Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Carcinoma, Renal Cell | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HLX17 (Experimental): Subjects will receive HLX17 (200 mg) on Day 1 of each 3-week cycle, until 12 months after the randomization (nearly 17 cycles) or investigator-assessed disease recurrence, death, initiation of new anti-tumor therapy, unacceptable drug toxicity, withdrawal of informed consent form, or study termination (whichever occurs first).
  Interventions: Drug: HLX17
- US-sourced Keytruda® (Active Comparator): Subjects will receive US-sourced Keytruda® (200 mg) on Day 1 of each 3-week cycle, for a total of 8 cycles (24 weeks). After 8 cycles, all subjects in the US-sourced Keytruda® group will receive HLX17 200 mg on Day 1 of each 3-week cycle until 12 months after the randomization (nearly 17 cycles) or investigator-assessed disease recurrence, death, initiation of new anti-tumor therapy, unacceptable drug toxicity, withdrawal of informed consent form, or study termination (whichever occurs first).
  Interventions: Drug: HLX17; Drug: US-sourced Keytruda®

INTERVENTIONS:
Drug: HLX17 — Subjects will receive HLX17 (200 mg) on Day 1 of each 3-week cycle
  Other Names: pembrolizumab
Drug: US-sourced Keytruda® — Subjects will receive US-sourced Keytruda® (200 mg) on Day 1 of each 3-week cycle
  Other Names: pembrolizumab
  Arms: US-sourced Keytruda®

SUMMARY:
This is a multicenter, randomized, double-blind, parallel-controlled phase I clinical study to evaluate the similarity in PK profile, efficacy, safety, and immunogenicity of HLX17 vs. US-sourced Keytruda® in patients with resected non-small cell lung cancer (NSCLC) or melanoma (MEL), or renal cell carcinoma (RCC).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have signed and dated an Institutional Review Board/Independent Ethics Committee (IRB/IEC) approved written informed consent form (ICF) in accordance with regulatory and institutional guidelines.
2. At least 18 years and no older than 70 years at the time of signing the ICF.
3. 18 kg/m2 ≤ body mass index (BMI) ≤ 30 kg/m2 and 50 kg ≤ body weight ≤ 85 kg.
4. The patient with one of the following resected solid tumors:

   * Stage IB (T2a ≥ 4 cm), II, or IIIA NSCLC patients after complete resection OR
   * Stage IIB, IIC, or III melanoma following complete resection OR
   * Renal cell carcinoma (RCC) at intermediate-high or high risk of recurrence following nephrectomy, or following nephrectomy and resection of metastatic lesions.
5. Have a performance status of 0 on the Eastern Cooperative Oncology Group (ECOG) Performance Status within 7 days prior to the first dose in this study.
6. Have a life expectancy of at least 12 weeks.
7. Have adequate organ function as indicated by the following laboratory values (no blood transfusions, or treatment with albumin, recombinant human thrombopoietin or colony-stimulating factor within 14 days prior to the first dose in this study)
8. Female patients must meet one of the following conditions:

   1. Menopause (defined as no menstruation for at least 1 year with no confirmed cause other than menopause), or
   2. Surgically sterilized (removal of the ovaries and/or uterus), or
   3. Fertile, but must:

      * be tested negative for serum/urine pregnancy test within 7 days prior to the randomization, and
      * agree to use contraception methods with an annual failure rate of < 1% or to remain abstinent (avoid heterosexual intercourse from signing the ICF to at least 6 months after the last dose of the study drug) (a contraceptive method with an annual failure rate of < 1% includes bilateral tubal ligation, male sterilization, correct use of hormonal contraceptives that can inhibit ovulation, hormone-releasing intrauterine devices and copper-containing intrauterine devices or condoms), and
      * not breastfeed
9. Male patients must: agree to remain abstinent (avoid heterosexual intercourse) or take contraception measures as follows: male patients with a pregnant partner or a partner of childbearing potential must remain abstinent or use condoms to prevent drug exposure to the embryo during study treatment and for at least 6 months after the last dose of study drug. Periodic abstinence (e.g., contraception based on calendar day, ovulatory phase, basal body temperature, or postovulatory phase) and external ejaculation are ineligible methods of contraception.

Exclusion Criteria:

1. Pregnant or lactating women.
2. History of illicit drug use or alcohol abuse within 12 months prior to randomization in the investigator's judgment.
3. Subjects with NSCLC have two synchronous primary non-small cell lung cancers or other histopathological types (such as mixed adenosquamous carcinoma, small cell lung cancer or neuroendocrine carcinoma).
4. Subjects with MEL have mucosal or ocular melanoma.
5. Subjects with RCC have pre-existing brain or bone metastatic lesions, or residual thrombus in the renal vein or vena cava after nephrectomy.
6. Subjects with other primary active malignancies within 5 years or at the same time prior to randomization.
7. Have received an organ or bone marrow transplantation prior to randomization or scheduled for transplantation during the study.
8. Presence of central nervous system (CNS) metastases and/or carcinomatous meningitis.
9. Symptomatic cerebrovascular disease or known myocardial infarction or poorly controlled arrhythmia (including QTc intervals ≥ 450 ms for males and ≥ 470 ms for females calculated by Fridericia's formula) within 6 months prior to randomization.
10. Chronic heart failure (Class III to IV based on NYHA classification) or an LVEF (left ventricular ejection fraction) assessed with the doppler echocardiography less than 50%.
11. Peripheral neuropathy greater than or equal to Grade 2 (CTCAE).
12. Known human immunodeficiency virus (HIV) infection (or positive anti-HIV during screening), or known Hepatitis B (or positive test for HBsAg or HBcAb and positive test for HBV-DNA during screening), or known Hepatitis C (or positive tests for HCV antibody and HCV-RNA during screening), or known Hepatitis B and C co-infection (or positive test for HBsAg or HBcAb and positive test for HCV antibody during screening), or active pulmonary tuberculosis within 6 months prior to randomization.
13. Known interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, and severe lung function abnormalities that may impede the investigators' diagnosis and management of drug-related pulmonary toxicity prior to screening.
14. Known severe allergic or anaphylactic reactions to pembrolizumab or any other monoclonal antibody or any components of the investigational medicinal products.
15. Known active or suspected autoimmune diseases. Patients with stable disease who do not require systemic immunosuppressive therapy may also participate.
16. Unstable hyperthyroidism or hypothyroidism at screening.
17. Have received live vaccines within 28 days prior to the first dose in this study (Inactivated viral vaccines for seasonal influenza are allowed).
18. Treatment with systemic corticosteroids (> 10 mg/day prednisone efficacy dosage) or other immunosuppressive drugs within 14 days prior to the first dose or during the study. However, subjects are allowed to be enrolled under the following conditions: in the absence of active autoimmune disease, subjects are allowed to use topical or inhaled steroids and adrenal hormone replacement therapy at dosages equivalent to ≤ 10 mg/day of prednisone efficacy.
19. Any active infection requiring systemic therapy within 1 month prior to the first dose in this study.
20. Subjects have planning to undergo surgical treatment during this clinical trial. Tumor puncture or incisional lymph node biopsy is allowed.
21. Have received pembrolizumab or any other immune checkpoints inhibitors (PD-1, PD-L1, CTLA4, etc.) before randomization.
22. Subjects have participated in a clinical study with another investigational medicinal product prior to randomization, and the interval between the current study and the previous study is too short: within 1 month prior to the first dose of the current study or within 5 half-lives of the previous investigational medicinal product (whichever is longer). Or planning to participate in a clinical study with another investigational medicinal product before completing all scheduled assessments in this clinical study.
23. Subjects have participated in a device clinical study within 1 month prior to screening, or are participating in another surgical or device clinical study at the time of screening, or plan to participate in another surgical or device clinical study during this clinical study.
24. The investigator has a clear reason to believe that participation in this study would be detrimental to the subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-03-27 (Estimated)

PRIMARY OUTCOMES:
AUC0-21d | rom time 0 to 21 days after the 1st dose (3 weeks)
  Area under the serum concentration-time curve from time 0 to 21 days (AUC0-21d) after the 1st dose
AUCss | from time 0 to 21 days after the 6th dose (18 weeks)
  Area under the serum concentration-time curve within a dosing interval at steady state (AUCss) after the 6th dose

SECONDARY OUTCOMES:
maximum serum drug concentration (Cmax), | up to 24 weeks
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
trough serum drug concentration at steady state (Ctrough,ss) | up to 24 weeks
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
maximum serum drug concentration at steady state (Cmax,ss) | up to 24 weeks
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
trough serum drug concentration (Ctrough) | up to 24 weeks
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
DFS | up to 12 months
  Defined as the time from randomization to tumor recurrence, the development of new tumor lesions, or death due to any reasons (whichever occur first).
Adverse events | From enrollment to the end of 90-day safety follow-up (up to 15 months)
  Adverse events (AEs) Serious adverse events (SAEs) Adverse events of special interest (AESIs) (including immune-related adverse events and infusion-related reactions)
Number of participants with abnormal vital signs | From enrollment to the end of 30-day safety follow-up (up to 13 months)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Number of participants with abnormal physical examination findings | From enrollment to the end of 30-day safety follow-up (up to 13 months)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Number of participants with abnormal Laboratory tests results (hematology, serum chemistry, thyroid function, coagulation function, and myocardial markers) | From enrollment to the end of 30-day safety follow-up (up to 13 months)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Number of participants with abnormal 12-lead ECG readings | From enrollment to the end of 30-day safety follow-up (up to 13 months)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Immunogenicity endpoint | up to 24 weeks
  Incidence of anti-drug antibody (ADA) and/or neutralizing antibody (NAb)

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial Cancer Hospital, Hunan, Changsha, China

IPD SHARING:
Plan to Share IPD: No